CLINICAL TRIAL: NCT00971841
Title: Rollover Study of Weekly Paclitaxel (BMS-181339) in Patients With Advanced or Recurrent Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA139-557
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Results first posted 2013-07-19 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Paclitaxel; BMS 181339

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel (Experimental): One hour intravenous infusion on Days 1, 8, 15, 22, 29, 36, followed by 1 week of rest (6 weeks on, 1 week off). One treatment course consists of 49 days. Day 1 dose same level as last dose of original Study CA139-540 (100mg/m2, 80 mg/m2, or 60 mg/m2). Treatment to continue until disease progression or unacceptable toxicity apparent.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel
  Other Names: Taxol; BMS-181339

SUMMARY:
The purpose of this study is to provide access to paclitaxel therapy to subjects with advanced or recurrent esophageal cancer who have completed the previous Phase 2 study (CA139-540) and who should continue on therapy with paclitaxel as assessed by the treating investigator(s). To evaluate the severity of observed adverse reactions in treated subjects for assessment of long-term safety.

ELIGIBILITY:
Subjects with advanced or recurrent esophageal cancer who have completed the previous late Phase 2 study (CA139-540) and for who continued therapy with paclitaxel would be beneficial as deemed by the investigator(s).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Original Study CA139-540 (NCT 00344552) at Dr. K. Kato National Cancer Center Hospital in Tokyo, Japan, closed in 2008 and one participant rolled over into Study CA139-557.
Pre-assignment Details: To be enrolled in Study CA139-557, participants with advanced or recurrent esophageal cancer must have completed original Study CA139-540 (NCT 00344552) and investigator(s) deemed that continuing treatment with paclitaxel would benefit the participant.
Groups:
- Paclitaxel: Paclitaxel dosed at the same dose level as last dose received in original study (100 mg/m^2, 80 mg/m^2, or 60 mg/m^2) and administered on Days 1, 8, 15, 22, 29, 36, followed by 1 week of rest (6 weeks on, 1 week off). One treatment course consisted of 49 days total.
Period: Overall Study
Arm/Group | Paclitaxel
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Paclitaxel: Paclitaxel dosed at the same dose level as last dose received in original Study CA139-540 (NCT 00344552)and administered on Days 1, 8, 15, 22, 29, 36, followed by 1 week of rest. One treatment course consisted of 49 days total.
Arm/Group | Paclitaxel
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 47 (NA) — Only one participant, therefore no standard deviation available.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  Japan | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events (AEs) Per Participant
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. Severity of the adverse event was judged and graded according to the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 2.0.
Time Frame: Weekly Day 1 to 4 years
Population: Only one participant enrolled in the study so all results represent one participant.
Measure: Number; unit: adverse events
Groups:
- Paclitaxel: Paclitaxel dosed weekly (6 weeks on, 1 week off).
Arm/Group | Paclitaxel
Number analyzed (Participants) | 1
adverse events | 32

2. Secondary Outcome: Number of Participants With Complete Response to Tumor
Description: Tumor measured/evaluated via imaging and assessed according to the Response Evaluation Criteria in Solid Tumor (RECIST) version 1.0 wherein complete response is disappearance of all target lesions; partial response is 30% decrease in the sum of the longest diameter of target lesions; progressive disease is 20% increase in the sum of the longest diameter of target lesions, and stable disease is small changes that do not meet above criteria. The baseline assessment was done prior to the first administration of drug in the original Study CA139-540 (NCT 00344552).
Time Frame: Every 7 weeks Day 1 to 4 years
Population: Only one participant enrolled so results are for one participant.
Measure: Number; unit: participants
Arm/Group | Paclitaxel
Number analyzed (Participants) | 1
participants | 1

ADVERSE EVENTS:
Time Frame: 4 years (4 March 2008 to 24 March 2012)
Arm/Group | Paclitaxel
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel (N=1)
neutrophil count decrease (Investigations) | 1 (44) — 16 events were Grade 1, 26 events were Grade 2 and 2 events were Grade 3
alopecia (Skin and subcutaneous tissue disorders) | 1 (30) — 29 events were Grade 1; 1 event was Grade 2
back pain (Musculoskeletal and connective tissue disorders) | 1 (13) — 11 events were Grade 1; 2 events were Grade 2
blood pressure increased (Investigations) | 1 (1) — 1 event Grade 1
chills (General disorders) | 1 (1) — Grade 1 event
contusion (Injury, poisoning and procedural complications) | 1 (2) — Grade 1 events
cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) — Grade 1 events
cystitis (Infections and infestations) | 1 (2) — one event Grade 1; one event Grade 2
decreased appetite (Metabolism and nutrition disorders) | 1 (2) — Grade 1 events
dizziness (Nervous system disorders) | 1 (11) — Grade 1 events
dry skin (Skin and subcutaneous tissue disorders) | 1 (3) — Grade 1 events
dysgeusia (Nervous system disorders) | 1 (1) — Grade 2 event
dysphagia (Gastrointestinal disorders) | 1 (2) — Grade 1 events
eczema (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 1 event
fatigue (General disorders) | 1 (2) — Grade 1 events
gingivitis (Gastrointestinal disorders) | 1 (3) — one Grade 1 event; two Grade 2 events
glucose urine present (Investigations) | 1 (2) — Grade 2 events
hemoglobin decreased (Investigations) | 1 (31) — One event Grade 1; 30 events Grade 2
herpes zoster (Infections and infestations) | 1 (2) — One Grade 1 event; one Grade 2 event
hypoesthesia (Nervous system disorders) | 1 (30) — 29 Grade 1 events; 1 Grade 2 event
malaise (General disorders) | 1 (6) — Five were Grade 1 events; one event was Grade 2
muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (12) — Grade 1 events
nasopharyngitis (Infections and infestations) | 1 (7) — Five events were Grade 1; 2 events were Grade 2
Nausea (Gastrointestinal disorders) | 1 (2) — Grade 1 events
edema (General disorders) | 1 (28) — 19 Grade 1 events; 9 Grade 2 events
periodontitis (Gastrointestinal disorders) | 1 (1) — Grade 1 event
peripheral motor neuropathy (Nervous system disorders) | 1 (4) — Grade 1 events
pharyngitis (Infections and infestations) | 1 (1) — Grade 2 event
protein urine present (Investigations) | 1 (2) — One Grade 1 event; one Grade 2 event
pyrexia (General disorders) | 1 (3) — Grade 1 events
weight decreased (Investigations) | 1 (5) — Grade 1 events
white blood cell count decreased (Investigations) | 1 (42) — 11 Grade 1 events; 31 Grade 2 events

LIMITATIONS AND CAVEATS:
Upon completion of Study CA139-540 (NCT 00344552), one subject (who had received 7 courses paclitaxel) rolled over into Study CA139-557. During four years in Study CA139-557, subject received an additional 30 courses of paclitaxel.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.